CLINICAL TRIAL: NCT03312413
Title: Efficacy of Dexmedetomidine for Cough Suppression During Anesthetic Emergence in Patients Undergoing Thyroid Surgery: A Randomized, Double Blinded, Controlled Trial
Brief Title: Efficacy of Dexmedetomidine for Cough Suppression in Patients Undergoing Thyroid Surgery
Acronym: EDCSTS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, clinical professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYYY2017
Record Dates: First submitted 2017-09-04; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia Complication
Keywords: dexmedetomidine; coughing during anesthetic emergence; thyroid surgery
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dexmedetomidine low dose group (Experimental): Patients in this group are received dexmedetomidine hydrochloride iv infusion of 0.2μg·kg-1·h-1 from incision to 20-30 minutes before the end of surgery
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Dexmedetomidine median dose group (Experimental): Patients in this group are received dexmedetomidine hydrochloride iv infusion of 0.5μg·kg-1·h-1 from incision to 20-30 minutes before the end of surgery
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Dexmedetomidine high dose group (Experimental): Patients in this group are received dexmedetomidine hydrochloride iv infusion of 0.7μg·kg-1·h-1 from incision to 20-30 minutes before the end of surgery
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Control group (normal saline group) (Placebo Comparator): Patients in this group are received saline iv infusion of 5mL·h-1 from incision to 20-30 minutes before the end of surgery
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine Hydrochloride 0.2 μg·kg-1·h-will be administered to participants by intravenous infusion from incision to 20-30 minutes before the end of surgery
  Arms: Dexmedetomidine low dose group
Drug: Normal Saline — Normal saline 0.5 mL·h-1 will be administered to participants by intravenous infusion from incision to 20-30 minutes before the end of surgery
  Arms: Control group (normal saline group)
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine Hydrochloride 0.5 μg·kg-1·h-1 will be administered to participants by intravenous infusion from incision to 20-30 minutes before the end of surgery
  Arms: Dexmedetomidine median dose group
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine Hydrochloride 0.7 μg·kg-1·h-1 will be administered to participants by intravenous infusion from incision to 20-30 minutes before the end of surgery
  Arms: Dexmedetomidine high dose group

SUMMARY:
Maintenance of a remifentanil infusion during anesthetic emergence has been reported to decrease the incidence of coughing and thereby help to ensure a smooth emergence. It may, however, cause respiratory depression and possibly delay emergence. The purpose of this study was to investigate the effect of different dose of dexmedetomidine infusion on cough suppression during emergence from general anesthesia in patients undergoing thyroid surgery.

American Society of Anesthesiologists physical status I-II adults undergoing elective thyroidectomy under general anesthesia are recruited and randomly allocated to receive dexmedetomidine iv infusion of 0.2μg·kg-1·h-1 (Group D1, n = 100), 0.5μg·kg-1·h-1 (Group D2, n = 100), 0.7μg·kg-1·h-1 (Group D3, n = 100) or saline (Group C, n = 100). Primary outcome is the incidence of coughing during emergence. Second outcomes include severity of coughing, which is assessed using a four-point scale; Ramsay score, Bruggrmann comfort scale score, VAS pain score are recorded. The respiratory rate (RR), heart rate (HR), and mean arterial pressure are also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. 30Kg/m2 ≥ BMI > 18Kg/m2;
2. undergoing general anesthesia;
3. ASA physical status I and II
4. undergoing elective thyroid surgery.

Exclusion Criteria:

1. hyperthyroidism;
2. preoperative bradycardia;
3. liver function impairment;
4. renal function impairment;
5. heart function failure;
6. history of asthma or COPD;
7. history of diabetes;
8. cognition function impairment;
9. pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of coughing during anesthetic emergence | within 10 minutes after endotracheal extubation
  incidence of coughing within 10 minutes after extubation

SECONDARY OUTCOMES:
Ccoughing on a four-point scale during anesthetic emergence | within 10 minutes after endotracheal extubation
  Evaluate the severity of coughing within 10 minutes after extubation by a four-point scale
Ramsay score during anesthetic emergence | within 30 minutes after endotracheal extubation
  Ramsay score 1min, 5min, 10min, and 30min after extubation
Bruggrmann comfort scale score | within 24 hrs after endotracheal extubation
  Bruggrmann comfort scale score 30min and 24 hrs after extubation
VAS pain score | within 48 hrs after endotracheal extubation
  VAS pain score 30min, 24 hrs and 48 hrs after extubation
Respiratory rate (RR) | within 30min after endotracheal extubation
  Respiratory rate 1min, 5min, 10min, and 30min after extubation
Heart rate | within 30 minutes after endotracheal extubation
  Heart rate 1min, 5min, 10min, and 30min after extubation
mean arterial pressure | within 30 minutes after endotracheal extubation
  Mean arterial pressure 1min, 5min, 10min, and 30min after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- China,Chongqing The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No